CLINICAL TRIAL: NCT04750928
Title: A Phase 0/I/II Study of the Cyclin-Dependent Kinase(CDK)4/6 Inhibitor Abemaciclib for Neurofibromatosis Type 1 (NF1) Related Atypical Neurofibromas
Brief Title: Cyclin-Dependent Kinase (CDK)4/6 Inhibitor Abemaciclib for Neurofibromatosis Type I (NF1) Related Atypical Neurofibromas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 210011; 21-C-0011
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12-04

CONDITIONS: Neurofibromatosis 1
Keywords: Kinase Inhibitor; distinct nodular lesion; genomic alteration
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — abemaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I Dose Escalation (Experimental): Abemaciclib orally twice daily at escalating doses to determine the MTD/RP2D
  Interventions: Drug: Abemaciclib
- 2/ Phase II Objective Response Rate (Experimental): Abemaciclib orally twice daily at the RP2D
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib is to be administered orally on Days 1 through 28 of each 28-day cycle

SUMMARY:
Background:

NF1 is a genetic disease that causes tumors called atypical neurofibromas. These tumors, which arise from nerves, can cause serious medical problems. The only treatment is surgery. Researchers want to see if a drug called abemaciclib can help.

Objective:

To find a safe, tolerable dose of abemaciclib for treating atypical neurofibromas.

Eligibility:

People ages 12 and older who have NF1 and have one or more atypical neurofibromas that cannot or will not be removed with surgery

Design:

Participants will be screened with:

Medical history and physical exam

Blood, urine, and heart tests

MRI: Participants will lie in a machine that takes pictures of the body. A padding or coil will be placed around their head. They may have a contrast agent injected into a vein.

Biopsy sample: A small piece of tumor will be removed using a large needle.

Participants will have frequent visits during the study. These will include repeats of the screening tests as well as the following:

PET scan: Participants will lie in a machine that takes pictures of the body. They will have a contrast agent injected into their arm.

Questionnaires about the effects of abemaciclib on pain and quality of life

Possible photographs of tumors

Participants will take abemaciclib capsules orally twice daily in 28-day cycles. They will take the drug for up to 2 years. Some may be able to take it for longer.

Participants will have a follow-up visit about 30 days after their last dose of the study drug. Then they will have visits every 3 months for 1 year.

DETAILED DESCRIPTION:
Background:

* Neurofibromatosis type 1 (NF1) is a genetic tumor predisposition syndrome (incidence of 1:3000), which results in the development of progressive tumor and non-tumor manifestations, the majority of which have no effective medical therapies. 25-50% of individuals with neurofibromatosis type 1 (NF1) develop histologically benign plexiform neurofibromas (PN), which can cause substantial morbidity. Recently, the POB identified that MEK inhibitors cause shrinkage of the majority of PN and that PN shrinkage is associated with clinical benefit.
* A natural history study of NF1 at the NCI has gathered comprehensive imaging information using longitudinal whole-body MRI with volumetric measurements. By this approach, distinct nodular lesions (DNL) were identified, many of which are atypical neurofibromas (ANF) based on pathology review.
* The NCI POB and others have described ANF as precursor lesions for aggressive soft tissue sarcomas called malignant peripheral nerve sheath tumors (MPNST), which show poor response to chemotherapy and have poor survival. Of note, ANF appear to be less responsive to treatment with MEK inhibitors indicating a different biology.
* Exome sequencing of 16 ANF resected at the National Cancer Institute, Pediatric Oncology Branch (NCI POB) and Belgium revealed that 90% of the cases had heterozygous loss of CDKN2A/B as the only new somatic change in addition to biallelic NF1 deletion, consistent with prior reports. These results demonstrate that transformation of NF1 nerve tumors may genetically proceed through the premalignant ANF by a common mechanism that might be a point of intervention.
* CDKN2A is the primary inhibitory brake on CDK4/6 driven signaling and is commonly deleted in glioblastoma, pancreas, bladder, breast and prostate cancer. The specific CDK4/6 inhibitor, abemaciclib, has FDA approval for the treatment of metastatic breast cancer.
* ANF is a prototypic premalignant lesion for testing experimental intervention, as these lesions are at risk for transformation, and share a common potentially druggable genomic alteration (CDKN2A/B deletion). We propose a clinical trial of abemaciclib in children and adults with NF1 and unresectable ANF.

Objectives:

* Phase 0: To determine the pharmacodynamic effect of 7-10 days of abemaciclib treatment prior to tumor resection on levels of phosphorylated Retinoblastoma (pRb)
* Phase I: To determine the recommended Phase II dose (RP2D) of abemaciclib in participants with NF1 and a measurable ANF
* Phase II: To determine the objective response rate (ORR) in the target ANF; complete and partial response (CR + PR), response determined by volumetric MRI analysis (>=20% volume reduction) compared to baseline

Eligibility:

* Participants must be at least 12 years of age with a diagnosis of NF1 with associated agerelated requirements as follows:

  * Willingness of participants >= 12 years old and <18 years old to undergo pretreatment percutaneous biopsy of ANF if deemed feasible with minimal morbidity
  * Willingness of participants >=18 years old to undergo pre-treatment and ontreatment percutaneous biopsy of ANF if deemed feasible with minimal morbidity
* Phase 0 Only:

  * Age >= 18 years old
  * Presence of >= 1 measurable ANF (biopsy confirmed) for which surgical removal at the NIH would not likely cause significant morbidity and is clinically indicated
* Phase I/II Only:

  --Presence of >= 1 measurable ANF (biopsy confirmed) for which surgical removal could cause significant morbidity OR for which participant is unwilling to undergo surgical resection OR the presence of more than one distinct nodular lesion (DNL) including at least 1 biopsy proven ANF
* For participants of all ages with ANF who cannot be safely biopsied with minimal morbidity, biopsy requirement to be performed at NIH Clinical Center will be waived from eligibility criteria. In this case, review of available archival tissue by NIH Pathology will be necessary to confirm diagnosis of ANF, which is mandatory for eligibility.

Design:

* This is a Phase 0/I/II non-randomized, open label, single institution study of the CDK4/6 inhibitor, abemaciclib, in children and adults with NF1 and a measurable ANF or with multiple ANF/DNL.
* The accrual ceiling will be set at 55 eligible participants (to include participants who are screened but found to not be eligible to undergo treatment).
* Phase 0: For participants with a biopsy-proven ANF that can be removed without significant anticipated clinical morbidity and where resection of the ANF is clinically indicated

  * Participants will receive abemaciclib at the same dose level and schedule as the Phase I/II portion at the time of enrollment for at least 7 days and no more than 10 days immediately prior to tumor resection
  * Tumor will be fully resected as per clinical care and participants will discontinue study drug
  * Participants will be followed for 30 days post-treatment or until resolution to <=grade 1 of any abemaciclib-related adverse events
  * The phase 0 study will have a 2-stage design with 3 participants in the first stage and an expansion to a total of 5 participants if at least one of the initial 3 participants achieves a pharmacodynamic response
* Phase I/II: For participants with a biopsy-proven ANF for which surgical removal could cause significant morbidity OR for which participant is unwilling to undergo surgical resection OR the presence of more than one distinct nodular lesion (DNL)

  * Primarily because the tolerability of investigational agents may differ between the NF1 population and non-NF1 population and secondarily because abemaciclib has not been evaluated in children to date, there will be a limited dose finding phase.
  * During the Phase 1 portion of the trial, the first 6 participants enrolled will be treated at 75% of the adult recommended Phase II dose (ARP2D; 150mg PO BID) of abemaciclib used in participants with malignancies, in a 28-day cycle. For participants < 18 years of age, dosing will be based on body surface area (BSA).
  * Cohorts of up to 6 participants will be enrolled, with dose adjustment depending on dose-limiting toxicities (DLT) until the maximum tolerated dose (MTD)/ recommended Phase II dose (RP2D) is established.
  * The Phase II trial is a Simon minimax two-stage trial design. An observed response rate of approximately 30% or greater would be considered desirable. The first stage of the Phase II portion of the trial will enroll 15 evaluable participants; if 0 to 2 of the 15 have a PR or CR, then no further participants will be accrued. If 3 or more of the 15 participants have a PR or CR, then accrual would continue until a total of 21 evaluable participants have been enrolled in phase II.
  * All participants will undergo careful toxicity monitoring. Restaging MRI for response will be performed pre-cycles 3 and 5, and then every 4 cycles for remainder of the first year.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All Participants
* Participants must have a clinical diagnosis of NF1, i.e., participants must have at least two of the diagnostic criteria for NF1 or a confirmed NF1 mutation from a CLIA-certified laboratory:

  * Six or more caf(SqrRoot)(Copyright)-au-lait macules (>= 0.5cm in prepubertal participants or >= 1.5 cm in post pubertal participants)
  * Freckling in axilla or groin
  * A neurofibroma or plexiform neurofibroma
  * Optic glioma
  * Two or more Lisch nodules
  * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
  * A first-degree relative with NF1
* Measurable disease: Participants must have at least one measurable ANF defined as a lesion of at least 3 centimeters (cm) measured in one dimension. Measurability and suitability for volumetric MRI analysis of the target ANF must be confirmed with the NCI POB prior to enrolling a participant. The target ANF will be defined as the clinically most relevant ANF, which has to be amenable to volumetric MRI analysis.
* Prior Therapies:

  * Since there is no standard effective chemotherapy for patients with NF1 and ANF, participants may be treated on this trial without having received prior medical therapy directed at their ANF.
  * Investigational agents/biologic therapies (not chemotherapy): Participants who have received previous investigational agents or biologic therapies are eligible for enrollment. At least 30 days or 5 half-lives must have elapsed since receiving medical therapy directed at any NF1 related tumor. Participants who received prior medical therapy for a NF1 related tumor manifestation must have recovered from the acute toxic effects of all prior therapy to grade 1 CTCAEv5 except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment before entering this study.
  * Chemotherapy agents: Participants who received chemotherapy must have recovered (CTCAE Grade <=1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to enrollment. A washout period of at least 28 days is required between last chemotherapy dose and enrollment (provided the participant did not receive radiotherapy).
  * Participants who received adjuvant radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. Participants who have received previous radiation therapy are eligible for enrollment. At least 6 weeks must have elapsed since the last radiation therapy and start of treatment. The only target ANF cannot have received radiation previously.
  * At least 28 days must have elapsed since any major surgeries, with evidence of good wound healing. Minimally invasive biopsies and central line placements are not considered major surgeries.
  * Participants who have received prior treatment with abemaciclib or another specific CDK4/6 inhibitor are not eligible for enrollment
* Adequate performance scale (Lansky/Karnofsky >=70%).
* Adequate organ function as defined below:

  --Hematologic Function: Participants must have an absolute neutrophil count >=1500/microliter, hemoglobin >=9 g/dL (transfusion independent, defined as not receiving blood transfusion unless related to trauma or surgeries), and platelets >=100,000/microliter (transfusion independent, defined as not receiving platelet transfusions unless related to trauma or surgeries)
* Hepatic Function: Participants must have bilirubin within 1.5 x the upper limit of normal for age, with the exception of those with Gilbert syndrome, and AST/ALT within <= 3 x upper limit of normal.
* Renal Function: Participants must have a creatinine clearance or radioisotope GFR >=60ml/min/1.73 m2 or a normal serum creatinine based on age, described in the table below.

  * Age (years) is >=12 and <=15 then Maximum Serum Creatinine (mg/dL) = 1.2
  * Age (years) >15 Maximum Serum Creatinine (mg/dL) = 1.5
  * Cardiac Function: Normal ejection fraction (ECHO or cardiac MRI) >= 53% (or the institutional normal; if a range is given then the upper value of the range will be used); QTC or QTcF <= 450 msec.
* Willingness to avoid grapefruit or grapefruit juice during abemaciclib administration
* Informed Consent: Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document. All participants or their legal guardians (if the participant is < 18 years old) must sign an IRB-approved document of informed consent to demonstrate their understanding of the investigational nature and the risks of this study before any protocol-related studies are performed. When appropriate, pediatric participants will be included in all discussions.
* Based on animal studies, the effects of abemaciclib can cause fetal harm. For these reasons, women of child-bearing potential and men must agree to use a highly effective contraceptive method during treatment and for at least 4 months after the last dose of abemaciclib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of abemaciclib administration

  * Woman participants of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first dose of abemaciclib.
  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>=12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Contraceptive methods may include intrauterine devices (IUD), or barrier method, a spermicidal agent should be added as a double barrier protection; abstinence is also acceptable.
  * Cases of pregnancy that occur during maternal exposures to abemaciclib should be reported. If a participant or spouse/partner is determined to be pregnant following abemaciclib initiation she must discontinue treatment immediately. Data on fetal outcomes and breastfeeding are to be collected for regulatory reporting and drug safety evaluation.
* Phase 0 Participants
* Presence of >= 1 measurable ANF (biopsy confirmed) for which surgical removal would not likely cause significant morbidity and is clinically indicated

NOTES: Definition of ANF. In addition, there will not be a requirement for confirmed CDKN2A/B deletion for study eligibility due to known biopsy sampling error and tumor heterogeneity.

* Age >= 18 years old
* Phase I/II Participants
* Presence of >= 1 measurable ANF (biopsy confirmed) for whom surgical removal could cause significant clinical morbidity OR for which participant is unwilling to undergo surgical resection OR the presence of more than one distinct nodular lesion (DNL) including at least 1 biopsy proven ANF

NOTES: Definition of ANF. In addition, there will not be a requirement for confirmed CDKN2A/B deletion for study eligibility due to known biopsy sampling error and tumor heterogeneity.

* Age >= 12 years old (no maximum age) with associated age-related requirements as follows:
* Age >= 12 years old with BSA >= 0.71 m2 and able to swallow whole tablets
* Willingness of participants >= 12 years old and <18 years old to undergo pretreatment percutaneous biopsy of ANF if deemed feasible with minimal morbidity
* Willingness of participants >= 18 years old to undergo pre-treatment and on-treatment percutaneous biopsy of ANF if deemed feasible with minimal morbidity

NOTE: For participants of all ages with ANF that cannot be safely biopsied with minimal morbidity, biopsy requirement to be performed at NIH Clinical Center will be waived from eligibility criteria. In this case, review of available archival tissue by NIH Pathology will be necessary to confirm diagnosis of ANF, which is mandatory for eligibility.

EXCLUSION CRITERIA:

* Pregnant women, or women who intend to become pregnant during the study, are excluded from this study because of the teratogenic effects of abemaciclib. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on study.
* May not have a NF1-related tumor such as optic pathway glioma or malignant peripheral nerve sheath tumor, which requires treatment with chemotherapy or surgery.
* Serious preexisting medical condition(s) that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel that would preclude adequate absorption, or preexisting Crohn s disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active bleeding diatheses or renal transplant, or psychiatric illness/social situations that would limit compliance with study requirements.
* Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Active bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Participants with HIV who have adequate CD4 counts and who have no requirement for antiviral therapy will be eligible.

NOTE:Screening is not required for enrollment.

* Participants with interstitial lung disease
* Requires treatment with strong CYP3A inhibitors or inducers
* Inability to swallow tablets, since tablets cannot be crushed or broken.
* Inability to undergo MRI and/or contraindication for MRI examinations following the MRI protocol. Prosthesis or orthopedic or dental braces that would interfere with volumetric analysis of target ANF on MRI.
* Refractory nausea and vomiting that would limit drug administration in the opinion of the Principal Investigator
* Known severe hypersensitivity to abemaciclib or any excipient of abemaciclib or history of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib
* Clinical judgment by the investigator that the participant should not participate in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
safety of abemaciclib in patients with NF1 and a measurable ANF | 30 days after treatment
  List of adverse event frequency

SECONDARY OUTCOMES:
Tolerability of abemaciclib on a prolonged dosing schedule | up to 2 years of treatment or until disease progression or unacceptable treatment-related toxicity
  Duration of treatment and adverse event types and frequency
Stable disease rate of target ANF | baseline through 30 days after treatment
  Proportion of patients that have progressive disease
Response rate of non-target ANF/DNL | at progression
  Changes in non-target ANF/DNL determined by volumetric MRI analysis
Effect of abemaciclib on CDK4/6 target inhibition | after Day 7 of Cycle 1
  Measurement of phosphorylated Retinoblastoma (pRB) in tumor biopsy samples
Effect of abemaciclib on ANF related pain and quality of life | baseline through 30 days after treatment
  Patient-Reported Outcome response
Abemaciclib pharmacokinetics and pharmacodynamic | 30 days after treatment
  Drug level in blood

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-C-0011.html